CLINICAL TRIAL: NCT03456843
Title: SIMCAP (Surgery in Metastatic Carcinoma of Prostate): Phase 2.5 Multi-Institution Randomized Prospective Clinical Trial Evaluating the Impact of Cytoreductive Radical Prostatectomy Combined With Best Systemic Therapy on Oncologic and Quality of Life Outcomes in Men With Newly Diagnosed Metastatic Prostate Cancer
Brief Title: Therapeutic Effect of Cytoreductive Radical Prostatectomy in Men With Newly Diagnosed Metastatic Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000031290; NCI-2018-00047 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 081707 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH); Pro20170001506 (Other: WIRB)
Record Dates: First submitted 2018-02-20; First posted 2018-03-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Stage IV Prostate Adenocarcinoma AJCC v7
MeSH Terms: interventions — Androgen Antagonists; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (ADT, docetaxel) (Experimental): Participants receive antiandrogen therapy with or without docetaxel at the discretion of the treating physician.
  Interventions: Drug: Antiandrogen Therapy; Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (ADT, radical prostatectomy, docetaxel) (Experimental): Participants receive antiandrogen therapy for at least 1 month, then undergo cytoreductive radical prostatectomy. Participants continue antiandrogen therapy and may receive docetaxel prior to surgery at the discretion of the treating physician.
  Interventions: Drug: Antiandrogen Therapy; Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: Antiandrogen Therapy — To demonstrate at least 30% improvement in FFS at 2 years after randomization with the power of 90% and error of 5% on a one-sided exponential MLE test.
  Other Names: ADT; Androgen Deprivation Therapy; Anti-androgen Therapy; Anti-androgen Treatment; Antiandrogen Treatment; Hormone Deprivation Therapy; Hormone-Deprivation Therapy
Drug: Docetaxel — To demonstrate at least 30% improvement in FFS at 2 years after randomization with the power of 90% and error of 5% on a one-sided exponential MLE test.
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Radical Prostatectomy — Undergo cytoreductive radical prostatectomy
  Other Names: Prostatovesiculectomy
  Arms: Arm II (ADT, radical prostatectomy, docetaxel)

SUMMARY:
This randomized phase II trial studies how well surgical removal of the prostate and antiandrogen therapy with or without docetaxel work in treating men with newly diagnosed prostate cancer that has spread to other places in the body. Androgens can cause the growth of prostate cancer cells. Antiandrogen therapy may lessen the amount of androgens made by the body. Drugs used in chemotherapy, such as docetaxel work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Surgery, antiandrogen therapy and docetaxel may work better in treating participants with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the clinical benefit of combining radical surgery cytoreductive radical prostatectomy (CRP) - with the best systemic therapy (BST) in men with newly diagnosed clinical metastatic prostate cancer (mPCa).

SECONDARY OBJECTIVES:

I. To determine the impact of CRP+BST on time to biochemical progression, cancer-specific survival, overall survival, complication rates, and quality of life (QOL) in patients with mPCa.

II. To determine the transcription levels of bone morphogenetic protein -6 (BMP-6) and transforming growth factor-beta (TGF-?).

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive antiandrogen therapy with or without docetaxel at the discretion of the treating physician.

ARM II: Participants receive antiandrogen therapy for at least 1 month, then undergo cytoreductive radical prostatectomy. Participants continue antiandrogen therapy and may receive docetaxel prior to surgery at the discretion of the treating physician.

After completion of study treatment, patients are followed up every 6 months from time of progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the prostate
* Evidence of metastasis by magnetic resonance imaging (MRI)/computed tomography (CT) scan, bone scan, or histologic confirmation
* Clinical stage M1a (distant lymph node positive), M1b (bone metastasis), or M1c (solid organ metastasis.
* If solitary lesion, metastasis confirmed with either biopsy or two independent imaging modalities (i.e. CT and PET [positron emission tomography], bone scan and MRI, modality at the discretion of the treating physician)
* No previous local therapy for prostate cancer (i.e prostate radiation, cryotherapy, etc.)
* Give informed consent
* Prostate deemed resectable by surgeon
* Plans to start or has already started antiandrogen therapy (ADT) no longer than 6 months prior to consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Hemoglobin (HgB) >= 9 g/dL compatible for surgery
* Platelets > 80,000/mcL compatible for surgery
* Aspartate aminotransferase (AST) =< 2x upper limit of normal (ULN) compatible for surgery
* Alanine aminotransferase (ALT) =< 2x upper limit of normal (ULN) compatible for surgery

Exclusion Criteria:

* Refuses to give informed consent
* Deemed to have unresectable disease by surgeon
* Received ADT for more than 6 months prior to consent
* Life expectancy of less than 6 months prior to consent
* Active spinal cord compression
* Deep vein thrombosis (DVT) / pulmonary embolism (PE) in the past 6 months prior to consent
* Previous local therapy for prostate cancer
* Patients who have chemotherapy or radiotherapy for non-prostate cancer related treatment within 3 weeks prior to consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS) | At 2 years
  Failure is defined as any one of the following events: PSA progression, clinical progression, radiographic progression, or death from prostate cancer. The % of men who fail within 2 years of randomization will be compare between the two groups using a one-sided log-rank test.

SECONDARY OUTCOMES:
Cancer-specific survival | Up to 2 years
Overall complication rate | Up to 2 years
Time to biochemical progression | Up to 2 years
Overall survival | Through study completion, a minimum of 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Kim, MD, Principal Investigator — Yale University
Locations (16):
- United States (7):
  - City of Hope, Duarte, California
  - University of California, Irvine, Irvine, California
  - University of Southern California, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Swedish Medical Services, Seattle, Washington
- Epworth Healthcare, East Melbourne, Australia, Australia
- Chinese University of Hong Kong, Hong Kong, China
- Japan (3):
  - Kindai University, Ōsaka-sayama, Osaka
  - Akita University, Akita
  - Juntendo University, Tokyo
- South Korea (3):
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Samsung Medical Center, Seoul
- National Taiwan University Hospital, Taipei, Taiwan